CLINICAL TRIAL: NCT03653390
Title: Efficacy and Mechanism of a Community Wellness Promotion Program for Middle-aged Adults Living With Long-term Physical Disability
Brief Title: A Community Wellness Program for Adults Living With Long-term Physical Disability
Acronym: EW-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ivan Molton, Professor, School of Medicine: Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00003931; R01NR016942-01 (NIH)
Record Dates: First submitted 2018-07-10; First posted 2018-08-31 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Physical Disability
Keywords: health promotion intervention; community participation; quality of life; middle age; multiple sclerosis; spinal cord injury; muscular dystrophy; post-polio syndrome
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries; Muscular Dystrophies; Postpoliomyelitis Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EnhanceWellness for Disability (EW-D) (Experimental): Up to 10 sessions of a telephone-based intervention delivered over a six-month period.
  Interventions: Behavioral: EnhanceWellness for Disability (EW-D)
- Wellness Education (Active Comparator): Eight 45-minute sessions of telephone-based wellness education delivered over a six-month period.
  Interventions: Behavioral: Wellness Education
- Control (No Intervention): Participant continues with their lives as they normally would.

INTERVENTIONS:
Behavioral: EnhanceWellness for Disability (EW-D) — Participants work one-on-one with the study Wellness Coach to identify health self-management problems, consider options, develop goals and an action plan, and make adjustments to that plan over time.
  Arms: EnhanceWellness for Disability (EW-D)
Behavioral: Wellness Education — Sessions will cover: (1) blood pressure management; (2) smoking cessation; (3) cancer screening; (4) regulation of blood glucose; (5) decreasing LDL cholesterol; (6) physical activity; (7) bone, joint, and muscle health; and (8) immunizations.
  Arms: Wellness Education

SUMMARY:
For people living with long-term physical disabilities, such as spinal cord injury or multiple sclerosis, middle-age (45-64) is a period of great vulnerability for losses in function and participation. There is an urgent need to develop and test interventions that can be delivered through existing community service agencies to help these people maximize their community participation and quality of life. This research will test the efficacy of one such intervention in a community trial and, thereby, contribute to our understanding of the intervention's effectiveness and mechanisms of action.

DETAILED DESCRIPTION:
Middle-age (45-64) is a time of health vulnerability for millions of Americans. More than 50% of individuals in the U.S. will have two or more chronic conditions by age 60, contributing to increased risk of later disability. However, for individuals with long-term physical disabilities (LTPDs) such as spinal cord injury or multiple sclerosis, these risks are magnified. This vulnerable population is especially in need of interventions to promote community participation and improve disease self-management during midlife.

Over the past 5 years, our research team has adapted an evidence-based health promotion intervention designed for older adults to serve middle-aged and older adults with LTPD. The investigators now have a trial version of this intervention (called "EnhanceWellness for Disability"; EW-D) with promising findings in pilot testing, ready for a larger community trial. Through a new partnership with 3 regional Centers for Independent Living, the investigators can now test this program for people with LTPD in 14 counties in the Northwest U.S.A.

The broad, long-term aims of this study are to test the efficacy of this program relative to two control conditions (an attention-matched health education control and treatment as usual), in 600 community dwelling adults age 45-64 years with LTPD using modern outcome scales appropriate for people with LTPD. The primary outcome is the ability to participate in valued community activities. The investigators will seek to determine whether the intervention was effective and if so, what mechanisms of change drove the effect. In addition to self-report, the investigators will also collect objective measures of community activity via global positioning system (GPS) and travel diaries, in a randomly selected subset of 300 participants. This study's specific aims are as follows:

Specific Aim 1. To determine the efficacy of eight sessions of EW-D, relative to an attention control condition or treatment as usual, in middle-aged adults with LTPD. The primary outcome will be the self-reported ability to participate in valued community activities.

Specific Aim 2. To determine if observed intervention effects are due to (1) improved disease management self-efficacy, (2) decreased interference due to pain and fatigue, or (3) improvements in psychological resilience.

Secondary Analyses. To determine if 1) intervention effects are maintained at 12 months and 2) intervention effects can be detected in objective, GPS -based measures of activity (quantified as number of trips outside the home, time outside the home, area of travel, and activity in established categories). The investigators will also examine the potential moderating effects of biological sex on treatment response.

This approach is consistent with goals described in recent National Institute on Aging (NIA) and National Institute of Nursing Research (NINR) program announcements, including those calling for age-appropriate interventions to improve self-management of chronic conditions (PA 14-344) and those calling for prevention research for adults in midlife (PA-15-098). If hypotheses are confirmed, this work would support a program that could be used to promote health and wellness in both able-bodied older adults and middle-aged adults with LTPD, which would be novel to the field and could improve reach.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 64 years of age at screening (turning 65 years after screening is ok);
* Able to read, speak, and understand English;
* Has a self-reported physician's diagnosis of long-term physical disability defined as:

  * a medical condition affecting the muscular or neurologic systems (eg, muscular dystrophy, multiple sclerosis, post-polio syndrome or spinal cord injury), and the condition:
  * creates functional disability (impairment in at least one activity of daily living (ADL) or at least one instrumental activity of daily living (IADL), as indicated by the Expanded Functional Disability Scale)
  * was present before age 40 years
* Able to participate via telephone;
* Has a goal in mind if randomized to the EW-D intervention;
* Has not participated in the original EnhanceWellness intervention group.

Exclusion Criteria:

* Under 45 years of age or 65 or older at screening;
* Unable to read, speak, or understand English;
* Does not have a neurological or muscular condition affecting physical function (e.g., persons with low back pain and shoulder pain would be excluded);
* Does not have functional disability;
* Disability onset after age 40 years;
* Significant cognitive impairment as defined by the Six-Item Screener;
* Psychiatric condition or symptoms that would interfere with participation, specifically:

  * Current, active suicidal ideation with current intent to harm oneself, or
  * Current schizophrenia, psychosis, or mania
* Unable to participate via telephone;
* Does not have a goal if randomized to the EW-D intervention;
* Has participated in the original EnhanceWellness intervention group.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 516 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Molton, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators propose to make available to interested researchers a data file (de-identified to remove any variables from which it would be possible to identify any individual participant) any data used in a published article, at the time that it is accepted for publication. That is, at the request of an outside researcher, the investigators will create and share a data file that includes all of the variables used in the published article and a list of the variables in the data file (along with their variable labels). Any investigators who request these data will receive (1) a copy of the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) a data set.
Time Frame: Data will become available after the main study results are published.
Access Criteria: Although any shared data will be stripped of identifiers prior to release, given the very specific nature of the study sample (middle-aged adults with disabilities) it is possible that those who access this data could potentially identify subjects with unusual characteristics or combinations of unusual characteristics. Therefore, the investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment and prior to group assignment, participants complete the baseline survey. Because participants have the option to withdraw at any time, some may choose to withdraw or are lost to follow up prior to randomization.
Groups:
- Wellness Education: Eight sessions of telephone-based wellness education delivered over a six-month period.
  Wellness Education: Sessions will cover: (1) blood pressure management; (2) smoking cessation; (3) cancer screening; (4) regulation of blood glucose; (5) decreasing LDL cholesterol; (6) physical activity; (7) bone, joint, and muscle health; and (8) immunizations.
Period: Overall Study
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Started | 183 | 159 | 163
3 Month Survey | 165 | 152 | 159
7 Month Survey | 165 | 150 | 156
Completed | 163 | 150 | 155
Not Completed | 20 | 9 | 8
Not completed — Lost to Follow-up | 12 | 8 | 7
Not completed — Withdrawal by Subject | 6 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Paper Survey Lost | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control | Total
Number analyzed (Participants) | 183 | 159 | 163 | 505
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 183 | 159 | 163 | 505
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 37 | 42 | 35 | 114
  Female | 145 | 117 | 127 | 389
  Transgender | 0 | 0 | 0 | 0
  Not Listed | 0 | 0 | 0 | 0
  Prefer not to Answer | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White / Caucasian | 162 | 145 | 144 | 451
  Black / African American | 14 | 9 | 12 | 35
  American Indian / Alaska Native | 7 | 3 | 2 | 12
  Asian / Asian American | 4 | 3 | 4 | 11
  Hawaiian Native / Pacific Islander | 3 | 0 | 0 | 3
  Other (Race) | 3 | 2 | 4 | 9
  Unknown | 0 | 0 | 0 | 0
  Prefer not to Answer (Race) | 0 | 0 | 1 | 1
  Hispanic | 6 | 7 | 6 | 19
  Not Hispanic | 176 | 151 | 156 | 483
  Other (Ethnicity) | 1 | 1 | 0 | 2
  Prefer not to Answer (Hispanic) | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 182 | 158 | 161 | 501
  Canada | 1 | 1 | 2 | 4
PROMIS Ability to Participate in Social Roles & Activities v2.0 Short Form 8a [Mean (Standard Deviation); unit: T-score] — 50 indicates the population mean with a standard deviation of 10. Higher scores represent greater perceived ability to participate in social roles and activities.
  T-score | 41.16 (7.79) | 41.90 (6.39) | 41.77 (7.36) | 41.60 (7.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Ability to Participate in Community Activities From Baseline to 6 Months
Description: Change in perceived ability to participate in community activities from baseline to 6 months. Assessed via the Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities short form (APSR). Higher scores indicate better ability to participate in social activities (total score range: 8-40)
Time Frame: Change from baseline to 6 months
Population: All participants with a PROMIS APSR value at both baseline and 6 months were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 161 | 148 | 154
score on a scale | 2.49 (5.95) | 1.25 (5.58) | 0.09 (4.80)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p < 0.01, ANOVA; The ANOVA was conducted on the change scores from baseline to 6 months
Statistical Analysis 2: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education; Test type: Superiority; p = 0.11, Tukey's HSD test; This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -1.24, 95% CI 2-sided [-2.71 to 0.22] — Difference is calculated as Wellness Education - EnhanceWellness for Disability
Statistical Analysis 3: Comparison: EnhanceWellness for Disability (EW-D) vs Control; Test type: Superiority; p < 0.01, Tukey's HSD test; This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -2.40, 95% CI 2-sided [-3.85 to -0.95] — Difference is calculated as Control - EnhanceWellness for Disability
Statistical Analysis 4: Comparison: Wellness Education vs Control; Test type: Superiority; p = 0.16, Tukey's HSD test; This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -1.16, 95% CI 2-sided [-2.64 to 0.32] — Difference is calculated as Control - Wellness Education

2. Secondary Outcome: Change in Self-report of Confidence in Managing One's Chronic Illness (Disease Management Self-efficacy) From Baseline to 3 Months
Description: Change in confidence in managing chronic illness, measured via the University of Washington Self-Efficacy Scale. Higher score indicates better self-efficacy (total score range: 6-30)
Time Frame: Change from baseline to 3 months
Population: All participants with a University of Washington Self-Efficacy Scale value at both baseline and 3 months were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 165 | 153 | 159
score on a scale | 2.19 (7.95) | 0.01 (7.06) | -0.07 (6.16)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p < 0.01, ANOVA; The ANOVA was conducted on the change scores from baseline to 6 months
Statistical Analysis 2: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education; Test type: Superiority; p = 0.018, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -2.18, 95% CI 2-sided [-4.05 to -0.30] — Difference is calculated as Wellness Education - EnhanceWellness for Disability
Statistical Analysis 3: Comparison: EnhanceWellness for Disability (EW-D) vs Control; Test type: Superiority; p = 0.012, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -2.26, 95% CI 2-sided [-4.12 to -0.41] — Difference is calculated as Control - EnhanceWellness for Disability
Statistical Analysis 4: Comparison: Wellness Education vs Control; Test type: Superiority; p = 0.99, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -0.08, 95% CI 2-sided [-1.98 to 1.81] — Difference is calculated as Control - Wellness Education

3. Secondary Outcome: Change in Self-reported Interference Due to Pain From Baseline to 3 Months
Description: Change in self-report of interference due to pain from baseline to 3 months, assessed via the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) short form. Higher scores indicate more pain interference (total score range: 4-20)
Time Frame: Change from baseline to 3 months
Population: All participants with a PROMIS PI value at both baseline and 3 months were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 165 | 153 | 159
score on a scale | -1.22 (6.47) | -0.55 (6.70) | -0.23 (6.66)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.382, ANOVA; The ANOVA was conducted on the change scores from baseline to 3 months

4. Secondary Outcome: Change in Self-reported Interference Due to Fatigue From Baseline to 3 Months
Description: Change in self-report of interference due to fatigue, from baseline to 3 months, assessed via the Patient-Reported Outcomes Measurement Information System Fatigue Interference short form. Higher scores indicate more fatigue interference (total score range: 4-20)
Time Frame: Change from baseline to 3 months
Population: All participants with a PROMIS fatigue measure at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 164 | 153 | 158
score on a scale | -1.89 (6.81) | -1.09 (6.85) | -0.76 (6.26)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.29, ANOVA; The ANOVA was conducted on the change scores from baseline to 3 months

5. Secondary Outcome: Change in Psychological Resilience From Baseline to 3 Months
Description: Change in self-report of psychological resilience, assessed via the Connor-Davidson Resilience Scale 10-item short form. Higher score indicates more resilience (total score range: 0-40)
Time Frame: Change from baseline to 3 months
Population: All participants with a Connor-Davidson Resilience score at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 164 | 150 | 157
score on a scale | 0.44 (5.61) | 0.28 (4.62) | -0.77 (4.20)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.057, ANOVA; The ANOVA was conducted on the change scores from baseline to 3 months

6. Secondary Outcome: Change in Number of Trips Outside the Home From Baseline to 12 Months
Description: Change in the average number of trips per day outside the home based on GPS data
Time Frame: Change from baseline to 12 months
Population: All participants with GPS data at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: trips per day outside the home
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 40 | 47 | 50
trips per day outside the home | -0.25 (0.84) | -0.12 (0.48) | 0.03 (0.83)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.21, ANOVA; The ANOVA was conducted on the change in number of trips from baseline to 12 months

7. Secondary Outcome: Change in Radius of Gyration From Baseline to 12 Months
Description: Radius of Gyration refers to a metric of activity space or overall mobility distance, calculated by creating a shape representing the area of daily travel, with a central index point, based on GPS data.
Time Frame: Change from baseline to 12 months
Population: All participants with GPS data at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 44 | 50 | 51
meters | 6328 (25527) | 6598 (105587) | 19917 (154597)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.79, ANOVA; The ANOVA was conducted on the change in radius of gyration from baseline to 12 months

8. Secondary Outcome: Change in Number of Trips Outside the Home Containing "Social" Elements From Baseline to 12 Months
Description: Change in the average number of trips per day outside the home containing "social" elements based on GPS and travel log data
Time Frame: Change from baseline to 12 months
Population: All participants with an average trips per day outside the home containing social elements measure at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: social trips outside the home M per day
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 37 | 42 | 44
social trips outside the home M per day | -0.18 (0.49) | -0.10 (0.41) | 0.02 (0.72)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p = 0.26, ANOVA; The ANOVA was conducted on the change in number of trips from baseline to 12 months

9. Secondary Outcome: Change in Time Spent in Activities Outside the Home Containing Social Elements From Baseline to 12 Months
Description: Change in average time per day spent in activities outside the home containing social elements from baseline to 12 months based on GPS and travel log data
Time Frame: Change from baseline to 12 months
Population: All participants with an average time per day spent in activities outside the home containing social elements measure at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 37 | 43 | 46
minutes | -30.1 (96.0) | -58.8 (145.2) | 36.5 (127.9)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p < 0.01, ANOVA; The ANOVA was conducted on the change in minutes from baseline to 12 months
Statistical Analysis 2: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education; Test type: Superiority; p = 0.57, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -28.7, 95% CI 2-sided [-95.7 to 38.4] — Difference is calculated as Wellness Education - EnhanceWellness for Disability
Statistical Analysis 3: Comparison: EnhanceWellness for Disability (EW-D) vs Control; Test type: Superiority; p = 0.048, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = 66.6, 95% CI 2-sided [0.56 to 132.6] — Difference is calculated as Control - EnhanceWellness for Disability
Statistical Analysis 4: Comparison: Wellness Education vs Control; Test type: Superiority; p < 0.01, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = 95.3, 95% CI 2-sided [31.8 to 158.7] — Difference is calculated as Control - Wellness Education

10. Secondary Outcome: Change in Self-reported Ability to Participate in Community Activities From Baseline to 12 Months
Description: Change in self-reported ability to participate in community activities from baseline to 12 months. Assessed via the Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities short form (APSR). Higher scores indicate better ability to participate in social activities (total score range: 8-40)
Time Frame: Change from baseline to 12 months
Population: All participants with a PROMIS APSR value at both baseline and 12 months were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
Number analyzed (Participants) | 158 | 145 | 153
score on a scale | 2.89 (4.92) | 1.34 (5.12) | 0.74 (5.65)
Statistical Analysis 1: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education vs Control; Test type: Superiority; p < 0.01, ANOVA; The ANOVA was conducted on the change scores from baseline to 12 months
Statistical Analysis 2: Comparison: EnhanceWellness for Disability (EW-D) vs Wellness Education; Test type: Superiority; p = 0.028, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -1.55, 95% CI 2-sided [-2.97 to -0.13] — Difference is calculated as Wellness Education - EnhanceWellness for Disability
Statistical Analysis 3: Comparison: EnhanceWellness for Disability (EW-D) vs Control; Test type: Superiority; p < 0.01, Tukey's HSD test; Mean Difference (Net) = -2.15, 95% CI 2-sided [-3.55 to -0.75] — Difference is calculated as Control - EnhanceWellness for Disability
Statistical Analysis 4: Comparison: Wellness Education vs Control; Test type: Superiority; p = 0.59, Tukey's HSD test — This test inherently adjusts for multiple comparisons; Mean Difference (Net) = -0.60, 95% CI 2-sided [-2.03 to 0.83] — Difference is calculated as Control - Wellness Education

ADVERSE EVENTS:
Time Frame: 1 year
Description: Other Adverse Events collected through regular inquiry with participants including during baseline, 3 mo, 6 mo, and 12 mo survey as well as during telephone based sessions with interventionist for EW-D and CDC Education arms over 6 month treatment window. Number of events differs from number of participants due to some participants reporting the same adverse event (both term and organ system) during the course of the year long study (e.g. multiple falls from same participant).
Arm/Group | EnhanceWellness for Disability (EW-D) | Wellness Education | Control
All-Cause Mortality (participants affected / at risk) | 1/183 | 0/159 | 0/163
Serious Adverse Events (participants affected / at risk) | 12/183 | 13/159 | 3/163
Other Adverse Events (participants affected / at risk) | 45/183 | 9/159 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EnhanceWellness for Disability (EW-D) (N=183) | Wellness Education (N=159) | Control (N=163)
Adverse Drug Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Participant reported non-study related drug reaction that resulted in hospitalization
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fall/Fall Related Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Post Surgical Complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Pressure Wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal Cord Injury Complications (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Throat Abscess (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Unknown Health Problem (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Participant reported hospitalization without specifying cause or outcome and was lost to follow up before collecting relevant information.
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EnhanceWellness for Disability (EW-D) (N=183) | Wellness Education (N=159) | Control (N=163)
Fall/Fall Related Injury (Injury, poisoning and procedural complications) | 18 (23) | 4 (4) | 0 (0) — Participant reports circumstances not meeting criteria for serious adverse event
Other Injury (Injury, poisoning and procedural complications) | 17 (19) | 3 (3) | 0 (0) — Participant reported injury not related to fall.
Multiple Sclerosis Related Symptom or Relapse (Nervous system disorders) | 10 (10) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Majority of participant recruitment took place during global COVID 19 pandemic which conceivably could have influenced participant outcomes in ways that could not be measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03653390/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03653390/SAP_001.pdf
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03653390/ICF_002.pdf